CLINICAL TRIAL: NCT02882243
Title: Post Market Study on the Safety and Efficiency of FLXfit™ TLIF Interbody Fusion Device (Cage)
Brief Title: FLXfit Post Market Outcome Study Protocol
Acronym: TLIF
Status: Completed | Type: Observational
Sponsor: Foundation for Orthopaedic Research and Education (Other)
Collaborators: CoreLink, LLC (Unknown)
Responsible Party: Principal Investigator, Marc Weinstein, Principal Investigator, Foundation for Orthopaedic Research and Education
Other Study IDs: 20-CL-027
Record Dates: First submitted 2016-07-15; First posted 2016-08-29 (Estimated); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Degenerative Disc Disease Lumbar

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: FLXfit Cage for fusion — Evaluating patient outcomes and radiographic outcomes
  Other Names: Transforaminal Interbody Fusion

SUMMARY:
This investigation will provide safety and effectiveness information on the use of the FLXfit™ Cage. Data will be used for Post Market follow-up of the FLXfit™ system by evaluating:

* Safety as measured by the rate of serious operative and post-operative complications.
* Patients' quality of life, measured by health-related quality of life questionnaires up to 24 months following the procedure, as compared to patient's baseline.

DETAILED DESCRIPTION:
Interbody fusion in patients with degenerative disc disease (DDD) at one or two contiguous levels from L2 to S1. Patients may also have up to Grade I spondylolisthesis or retrolisthesis at the involved level(s). Patients should be skeletally mature and have completed six months of non-operative treatment

ELIGIBILITY:
Inclusion Criteria:

* Adult (age 18 - 70 years) patient (male or female) with the following conditions of the lumbar spine as confirmed by advanced imaging (CT or MRI), who is a candidate for primary spinal fusion procedure according to acceptable criteria for such medical conditions:

  * Degenerative disc disease
  * With up to Grade I spondylolisthesis
* Failure of at least 6 month conservative treatment BMI < 40.
* Patient to approve no pregnancy during the 24 months of study and no participation in other studies in parallel to this one.

Exclusion Criteria:

* This device is not intended for cervical spine use. PI may exclude patient from study

Contraindications include, but are not limited to:

* Infection, local to the operative site
* Signs of local inflammation,
* Fever or leukocytosis,
* Morbid obesity,
* Pregnancy,
* Mental illness,
* Any other condition which would preclude the potential benefit of spinal implant surgery, such as the presence of tumors or congenital abnormalities, fracture local to the operating site, elevation of segmentation rate unexplained by other diseases, elevation of white blood count (WBC), or a marked left shift in the WBC differential count,
* Suspected or documented allergy or intolerance to implant's materials,
* Any case not described in the indications,
* Any patient unwilling to cooperate with postoperative instructions.
* These devices must not be used for pediatric cases, nor where the patient still has general skeletal growth.
* Any case where the implant components selected for use would be too large or too small to achieve a successful result.
* Any patient having inadequate tissue coverage over the operative site or inadequate bone stock or quality.
* Any patient in which implant utilization would interfere with anatomical structures or expected physiological performance.
* Prior fusion at the level to be treated.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Up to 50 subjects participating in this post market study will be consecutively recruited from the Clinical Investigators standard patient populations.
  * The Principal Investigator is responsible for assessing the eligibility of their potential subjects.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-07; Primary Completion 2022-01 (Actual); Study Completion 2022-07 (Actual)

PRIMARY OUTCOMES:
Improvement in Oswestry Disability Index (ODI) score | Baseline, 6 week, 3 month, 6 month, 12 month, 24 month follow-up
  Oswestry Disability Index is a measure of disability due to back and leg pain

SECONDARY OUTCOMES:
Disc Height | at 6 months
  measurement of overall lumbar lordosis and segmental disc height

IPD SHARING:
Plan to Share IPD: Undecided
not at this time